CLINICAL TRIAL: NCT01708382
Title: Feasibility Study: Evaluation of the Ulthera® System for Lifting and Tightening of the Elbow Tissue - A Feasibility Study
Brief Title: Feasibility Study: Lifting and Tightening of the Elbows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-108
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy treatment on the elbows (Experimental): All enrolled subjects will receive one Ultherapy treatment to the elbows.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
Up to 20 subjects will be treated. Treated subjects will receive one Ulthera® treatment on the elbows. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, single-center, pilot clinical trial to evaluate the efficacy of the Ulthera® System to improve skin laxity above the elbows. Masked assessment of pre- and post-treatment photos will be performed. Global Aesthetic Improvement Scale scores and patient satisfaction questionnaires will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 21 to 65 years.
* Subject in good health.
* Mild to moderate skin laxity on the elbows.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1 and be willing and able to use an acceptable method of birth control

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Excessive subcutaneous fat around the elbows.
* Excessive skin laxity around the elbows.
* Significant scarring in areas to be treated.
* Significant open wounds or lesions in the area to be treated

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Overall improvement of skin laxity in the areas treated | 90 days post-treatment
  Determined by masked assessment analysis of photographs at 90 days post treatment compared to baseline.

SECONDARY OUTCOMES:
Aesthetic improvement | 90 and 180 days post-treatment
  GAIS scores will be obtained by the Investigator and subjects at all visits excluding baseline. Additionally, subject satisfaction questionnaires will also be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron K Rokhsar, MD, Principal Investigator — New York Cosmetic, Skin, and Laser Surgery Center
Locations (1):
- New York Cosmetic, Skin and Laser Surgery Center, New York, New York, United States